CLINICAL TRIAL: NCT02963363
Title: Feasibility Study of an Adapted Physical Activity (APA) for Breast Cancer Patients Treated by Neoadjuvant Chemotherapy and Targeted Therapy Against HER2
Brief Title: Adapted Physical Activity for Breast Cancer HER2 Positive Patient
Acronym: APACAN2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-A01344-47
Record Dates: First submitted 2016-11-07; First posted 2016-11-15 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: HER2 Positive Breast Cancer
Keywords: Breast cancer; HER2+; Adapted physical activity; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Home-Based Adapted Physical Activity intervention during neoadjuvant chemotherapy :
  150 minutes per week of aerobic and muscle strengthening exercises during 18 weeks
  Interventions: Other: Home-based Adapted Physical Activity

INTERVENTIONS:
Other: Home-based Adapted Physical Activity — Home-based adapted physical activity to attend progressively 150 minutes of physical activity per week at the end of neoadjuvant chemotherapy.
  5 times 30 minutes of walking + 3 times 30 minutes of muscle strengthening exercises per week during 18 weeks

SUMMARY:
The purpose of this study is to assess the feasibility of a home-based adapted physical activity during neoadjuvant chemotherapy for HER2+ breast cancer.

DETAILED DESCRIPTION:
After the assessment of their physical fitness, a home-based adapted physical activity program composed by aerobic and muscle strengthening exercises will be delivered to each patient. The aim of the intervention is to reach international recommendation in a progressive way during neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years old
* Patient with HER2 (Human Epidermal growth factor Receptor 2) positive breast cancer histologically proven, eligible for neoadjuvant chemotherapy and targeted therapy against HER-2
* Affiliation to the French social security scheme
* Patient who signed the participation consent before entering the trial
* Medical fitness certificate for sport

Exclusion Criteria:

* Diagnosis of a second malignancy in the past 5 years, with the exception of a basal cell skin cancer
* Metastatic cancer
* Karnofsky index ≤ 90%
* Men
* Pregnant women
* Significant psychiatric or neurological abnormality
* Patient deprived of liberty by a court or administrative
* Contraindication for physical activity
* Patient unable to complete questionnaires (language barrier)
* Participation in a clinical trial with the same objective

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Rate of patients reaching international physical activity recommendations for post-neoadjuvant chemotherapy assessment | Change from baseline (T0: before neoadjuvant chemotherapy) at the 5 months (T1: end of neoadjuvant chemotherapy)
  Time spent to physical activity and sedentariness will be evaluated by Recent Physical Activity Questionnaire (RPAQ)

SECONDARY OUTCOMES:
Longitudinal evolution of RPAQ score | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
Quality of life : Quality of Life Questionnaire-C30 | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
Asthenia : Multidimensional Fatigue Inventory-20 | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
Anthropometrics measurements | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
  BMI
Anthropometrics measurements | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
  Hip circumference (cm)
Physical capacity : six-minutes walking distance test | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
Physical capacity : Voluntary muscular strength | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
Physical capacity : VO2max | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
  This measure is optional
Lipid profile : total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
Ventricular ejection fraction assessed by echocardiography or cardiac scintigraphy | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
Changes of cancer treatment | At each cycle of neoadjuvant chemotherapy : every three weeks during 5 months
  frequency of dose reduction (%), of postponement (%) or of treatment discontinuation (%)
Assessment of physical activity level using a validated smartphone application (eMouveRecherche) | Before (T0) and at the end (T1 : + 5 months) of neoadjuvant chemotherapy + before (T2 : + 8 months) and at the end (T3 : 20 month) of targeted therapy
  Including sedentariness time

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, MD, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France

REFERENCES:
- [Derived] Ginzac A, Bernadach M, Molnar I, Duclos M, Thivat E, Durando X. Adapted Physical Activity for Breast Cancer Patients Treated with Neoadjuvant Chemotherapy and Trastuzumab Against HER2 (APACAN2): A Protocol for a Feasibility Study. Front Oncol. 2021 Dec 13;11:744609. doi: 10.3389/fonc.2021.744609. eCollection 2021. PMID 34966667